CLINICAL TRIAL: NCT06499207
Title: Advanced Coronary Plaque Morphology Assessment Using Photon-counting Detection and Invasive Coronary Imaging
Acronym: ACDC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Eva Steinacher, MD, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ACDC_2547
Record Dates: First submitted 2024-06-11; First posted 2024-07-12 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Coronary Artery Disease; Coronary Disease; PCI; Stent Restenosis
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Photon-counting detector computed tomography (PCD-CT) — Patients undergoing follow-up coronary angiography with IVI after percutaneous coronary intervention (PCI) as part of routine clinical practice will additionally receive coronary computed tomography angiography (CCTA) with PCD as part of this study.

SUMMARY:
This clinical trial aims to compare non-invasive photon-counting detector computed tomography (PCD-CT) with invasive intravascular imaging (IVI) for post-interventional follow-up in patients with coronary artery disease (CAD).

Participants will undergo post-interventional follow-up using both PCD-CT and coronary angiography with IVI. Researchers will test qualitative and quantitative PCD-CT results for non-inferiority to IVI regarding stent evaluation and detection of in-stent restenosis and plaque morphology.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* DES in proximal coronary vessel segments

Exclusion Criteria:

- Any conditions that may interfere with the safety or efficacy of CCTA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Quantitative comparison of PCD-CT and IVI in stent evaluation | Within 1 year
  Comparison of post-PCI minimal stent area, stent diameter, stent lumen visualization, coronary wall visualization
Qualitative comparison of PCD-CT and IVI in stent evaluation | Within 1 year
  Two experienced radiologists/cardiologists will independently rate image noise and stent artefacts (1 = inadequate; 5 = excellent)

SECONDARY OUTCOMES:
Quantitative comparison of PCD-CT and IVI for the evaluation of in-stent restenosis | Within 1 year
  Severity of stenosis: Calculation of the percentage (%) of lumen diameter and lumen are stenosis with the appropriate CCTA and IVI analysis software
Quantitative comparison of PCD-CT and IVI for the evaluation of plaque morphology | Within 1 year
  Plaque morphology: Characterization of plaque components using Hounsfield units (HU) with the appropriate CCTA and IVI analysis software
Qualitative comparison of PCD-CT and IVI for the evaluation of in-stent restenosis and plaque morphology | Within 1 year
  Two experienced radiologists/cardiologists will independently rate the visualization of in-stent restenosis and plaque morphology using a five-point scale (1 = inadequate; 5 = excellent)

IPD SHARING:
Plan to Share IPD: Undecided